CLINICAL TRIAL: NCT00157976
Title: A Phase III Randomized, Multicenter, Multinational, Double-Masked, Placebo-Controlled Study of Photrex (Rostaporfin) Photodynamic Therapy in the Treatment of Classic and Occult Subfoveal Choroidal Neovascularization Associated With AMD
Brief Title: Double-Masked Study of Photrex (Rostaporfin) Photodynamic Therapy in the Treatment of Age-Related Macular Degeneration
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miravant Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MRVT-920101-OPH005
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-11

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration; AMD; Visual Acuity
MeSH Terms: conditions — Macular Degeneration | interventions — tin etiopurpurin

INTERVENTIONS:
Drug: Photrex (rostaporfin)

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of rostaporfin (PHOTREX) photodynamic therapy (PDT) in the treatment of classic and occult subfoveal choroidal neovascularization (CNV) associated with age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

Patients with age greater than or equal to 50 years with at least one subfoveal CNV membrane secondary to AMD that can be demonstrated by fluorescein angiography.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660
Dates: Start 2005-09

PRIMARY OUTCOMES:
Visual Acuity

SECONDARY OUTCOMES:
Angiographic changes

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J. Snyder, PhD, Study Director — Miravant Pharmaceuticals
Locations (4):
- Multiple Investigators, Sofia, Bulgaria
- Multiple Investigators, Brno-Bohunice, Olomouc, Praha, Czechia
- Multiple Investigators, Warsaw, Bydgoszcz, Lubin, Poland
- Multiple Investigators, Bucharest, Romania